CLINICAL TRIAL: NCT03431259
Title: Does Inpatient Enrollment Into a Patient Communication App (Patient Gateway) Result in Improved Follow-up and Survey Completion Rates After Orthopaedic Trauma?
Brief Title: Inpatient Enrollment of Patient Portal App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marilyn Heng, Instructor in Orthopaedic Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017P001594
Record Dates: First submitted 2018-01-20; First posted 2018-02-13 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enrollment group (Experimental)
  Interventions: Other: Patient Gateway
- Information group (No Intervention)

INTERVENTIONS:
Other: Patient Gateway — Patients will be enrolled in the Patient Gateway app.
  Arms: Enrollment group

SUMMARY:
This study aims to determine if inpatient enrollment into a patient communication app improves clinic follow-up of orthopedic trauma patients and improves survey completion rates after orthopedic trauma.

DETAILED DESCRIPTION:
Follow-up in trauma is historically poor. As a result, outcomes from trauma are difficult to collect via surveys and are often significantly influenced by selection bias. Patient interaction apps like Patient Gateway are thought to facilitate greater participant involvement and adherence to treatment regimens. The investigators will explore if inpatient enrollment into Patient Gateway would improve clinic follow-up rates. Increasing follow-up rates could improve the quality of care delivered.

In addition, self-administered survey questionnaires are an important data collection tool in clinical practice, public health research and epidemiology. However, survey completion rates are typically poor in orthopaedic trauma.

With the evaluation of modern technology, electronic applications are being increasingly used in both hospital and personal settings. In outpatient clinics, questionnaires to measure outcomes and monitor quality of care are administered by staff members using hospital owned tablet devices. Recently, applications to complete these surveys on personal devices have been developed.

In a recent Cochrane review on the comparison of self-administered survey questionnaire responses collected using mobile apps versus other methods it was concluded that there are no data available on response rates. The investigators will attempt to address this question.

All Patient Gateway naïve patients aged 18 years or older able to consent for themselves and admitted to the hospital for an orthopedic condition with the need for outpatient follow-up will be invited to participate in this study. Exclusion criteria will be patients unable to consent for themselves, inability to communicate in English, and no possession of a smartphone.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the hospital for an orthopedic condition with the need for outpatient follow-up
* able to consent for themselves

Exclusion Criteria:

* unable to consent for themselves
* inability to communicate in English
* no possession of a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhashyam AR, Bansal M, McGovern MM, van der Vliet QMJ, Heng M. In-hospital Enrollment Into an Electronic Patient Portal Results in Improved Follow-up After Orthopedic Surgery: Cluster Randomized Controlled Trial. JMIR Perioper Med. 2022 Aug 11;5(1):e37148. doi: 10.2196/37148. PMID 35969452

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrollment Group: Patient Gateway: Patients will be enrolled in the Patient Gateway app with the assistance of a research coordinator as an inpatient.
- Information Group: Patients will be provided with information sheet only on how to enroll for Patient Gateway app.
Period: Overall Study
Arm/Group | Enrollment Group | Information Group
Started | 115 | 117
Completed | 113 | 116
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enrollment Group | Information Group | Total
Number analyzed (Participants) | 113 | 116 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (16) | 54.5 (16.7) | 53.5 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 55 | 115
  Male | 53 | 61 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Non-White race | 21 | 17 | 38
  Race: White/Caucasian race | 92 | 99 | 191
Median income by Zipcode [Median (Standard Deviation); unit: dollars] | 83221 (26358) | 80888 (27853) | 82039 (27091)
Injury vs Acute Infection [Count of Participants; unit: Participants]
  Injury or Acute Infection | 48 | 45 | 93
  Elective | 65 | 71 | 136
Admission Subspecialty [Count of Participants; unit: Participants]
  Joints | 37 | 38 | 75
  Oncology | 4 | 5 | 9
  Sports/Shoulder | 5 | 5 | 10
  Spine | 18 | 23 | 41
  Trauma | 49 | 45 | 94

OUTCOME MEASURES:

1. Primary Outcome: Return to Clinic
Description: The number of patients enrolled who return to clinic for a followup visit at 3 months postop. It will be a count and proportion of the occurrence of a patient returning to clinic for followup
Time Frame: 3 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Enrollment Group | Information Group
Number analyzed (Participants) | 113 | 116
Participants | 97 | 93
Statistical Analysis 1: Comparison: Enrollment Group vs Information Group; Test type: Superiority; p = .0574, Chi-squared
Statistical Analysis 2: Comparison: Enrollment Group vs Information Group; Test type: Superiority; p = 0.570, Chi-squared

2. Primary Outcome: Use of Any the Patient Gateway Portal at 3 Months
Description: The number of patients who used the patient gateway portal for any purpose at 3 months. This will be a count of participants.
Time Frame: 3 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Enrollment Group | Information Group
Number analyzed (Participants) | 113 | 116
Participants | 70 | 19

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Enrollment Group | Information Group
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/116
Other Adverse Events (participants affected / at risk) | 0/113 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT03431259/Prot_SAP_000.pdf